



### Oyster Point Pharma, Inc.

**Clinical Protocol: OPP-005:** 

A Single-Center, Randomized, Controlled, Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation (The IMPERIAL Study)



### Statistical Analysis Plan for Safety Data Version 1.0

Prepared

Date: July 1, 2020



### **Revision History**





### **Prepared by:**







### Contents

| 1 | S | Synopsis | 5 |
|----|-----|-------------------------------------------------|----|
| 2 | A | Abbreviations | 6 |
| 3 | Iı | ntroduction | 7 |
| 4 | S | Study Objective | 7 |
| 5 | S | Study Design | 7 |
| 6 | S | Sample Size Determination and Power Calculation | 7 |
| 7 | S | Statistical Analysis | 7 |
| | 7.1 | General Consideration | 8 |
| | 7.2 | Analysis Populations | 8 |
| | 7 | 7.2.1 Safety population | 8 |
| | 7.3 | Definition of Study Day | 8 |
| | 7.4 | Missing and Partial Data | 8 |
| | 7.5 | Protocol Deviations | 9 |
| | 7.6 | Subject Disposition | 9 |
| | 7.7 | Demographics and Baseline Characteristics | 10 |
| | 7.8 | Medical, Ocular and Dry Eye History | 10 |
| | 7.9 | Treatment Exposure | 10 |
| 8 | Iı | ntranasal Examination | 10 |
| 9 | S | Safety Analysis | 10 |
| | 9.1 | Adverse Events | 10 |
| | 9.2 | Prior and Concomitant Medications | 11 |
| Αį | per | ndix 1 Schedule of Visits and Measurements | 13 |
| Αį | per | ndix 2 Table of Contents | 14 |
| Αį | per | ndix 3 Tableshell | 16 |





### 1 Synopsis

| A Single-Center, Randomized, Controlled, Masked Clinical Trial to Evaluate the |
|---|
| Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation |
| (The IMPERIAL Study) |
| OPP-005 |
| OC-01 (varenicline) Nasal Spray: |
| • 1.2 mg/mL |
| The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo in simulating Goblet Cell and Meibomian Gland function in adult subjects with DED. |
| 45 subjects will be randomized in a 2:1 ratio to the two treatment groups. |
| • 1.2 mg/mL |
| Placebo (vehicle) |
| Subjects who passed screening at Visit 1 will be randomized and administered study |
| drug in office at Visit 2. |
| The sample size for this study is not based on statistical power considerations. |
| Safety Endpoint: |
| Adverse Events |
| The safety population will include all randomized subjects who received study drug. |
| Analysis on the safety population will group subjects according to the treatment actually received. |





### 2 Abbreviations

ΑE adverse event

CRF case report form DED dry eye disease

FDA Food and Drug Administration

HIPAA Health Information Portability and Accountability Act

IΒ Investigator's Brochure **ICF** informed consent form **IRB** institutional review board

Milligram mg mL Milliliter

SAE serious adverse event SAP Statistical Analysis Plan

SD Standard deviation

TEAE treatment-emergent adverse event





### 3 Introduction

This statistical analysis plan (SAP) contains the detailed technical specifications for the safety data only described in the OPP-005 protocol Amendment #4 (26 March 2019).

The reviewer can refer to the study protocol and the case report form (CRF) for details of study design, conduct and data collection. Specifications of tables and data listings are contained in a separate document.

The objective of this SAP is to evaluate the safety of OC-01 (varenicline) Nasal Spray as compared to placebo on incidence of treatment-emergent adverse event (TEAE) in adult participants with dry eye disease (DED).

If the analyses described in the protocols differ from those in this SAP, the methods of the SAP prevail.

### 4 Study Objective

The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo in simulating Goblet Cell and Meibomian Gland function in adult subjects with DED.

### 5 Study Design

Protocol OPP-005 is a Phase 2, single-center, randomized, masked, placebo-controlled study designed to evaluate the safety of OC-01 Nasal Spray as compared to in adult participants with DED. Approximately 45 subjects at least 18 years of age with a physicians' diagnosis of dry eye disease and meeting all other study eligibility criteria will be randomized to receive an application of OC-01 or placebo at a single visit.

Appendix 1 describes the detailed study visits, measurements, and dosing information.

### **6** Sample Size Determination and Power Calculation

The sample size for this study is not based on statistical power considerations. The study will randomize approximately 45 subjects in a 2:1 ratio to the two treatment groups. It is expected that approximately 30 subjects will be enrolled in the investigational treatment arm and 15 subjects will be enrolled in the placebo arm. It is expected that all 45 subjects will be enrolled.

### 7 Statistical Analysis





### 7.1 General Consideration

Descriptive and inferential statistics will be used to summarize results of Protocol OPP-005. Continuous variables will be summarized using the number of subjects (n), mean, SD, median, 25<sup>th</sup> and 75<sup>th</sup> percentiles, and minimum and maximum. Categorical variables will be summarized using frequency counts and percentages. Baseline measures will be defined as the last measure prior to the initiation of study treatment.

All summaries for safety data will be presented by treatment group. For the demographics and baseline characteristics, all summaries will be presented by treatment group. All collected data will be presented in listings which will be sorted by treatment, subject ID, and visit when it is appropriate. Summaries, data listings, and statistical analyses will be generated using SAS® Version 9.4 or higher.

### 7.2 Analysis Populations

### 7.2.1 Safety population

The safety population will include all randomized subjects who received study drug at Visit 2. Analysis of the safety population will group subjects according to the treatment actually received.

### 7.3 Definition of Study Day

Study Day = [Event date – Randomization date + 1] if after randomization [Event date – Randomization date] if before randomization

Note that with the definition above, days of "0" will not be used.

For subjects whose reference date is missing, the study day will also be categorized as missing.

### 7.4 Missing and Partial Data





For all other cases, set date to date of first dose.

### Adverse event end date

If year is present and month and day are missing or year and day are present and month is missing, set end month and day to December 31.

If month and year are present and day is missing, set the day to last day of the month.

If fatal event, date is set to minimum of imputed end date and death date.

For all other cases, set date to missing.

For summaries that present distribution of time expressed in weeks and months, weeks will be defined as days divided by 7 and months as days divided by 30.4375.

### 7.5 Protocol Deviations

Important protocol deviations will be summarized by randomized treatment group.

### 7.6 Subject Disposition

The number and percentage of subjects randomized and included in analysis population will be summarized by treatment and overall.

The number of all subjects who completed the study and reasons for discontinuation will be summarized by treatment group and overall. The Case Report Form (CRF) lists the following reasons why subjects may discontinue study:

• Non-fatal adverse event (AE)





- Protocol violation
- Lost to follow-up
- Pregnancy
- Physician decision
- Subject non-compliance
- Death
- Study terminated by sponsor
- Withdrawal by subject
- Other reasons

### 7.7 Demographics and Baseline Characteristics

Demographic and baseline characteristics for safety population will be summarized using descriptive statistics by treatment group.

Continuous demographic and baseline variable includes age; categorical variables include gender, ethnicity, and race.

### 7.8 Medical, Ocular and Dry Eye History

Medical history terms and ocular history terms will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.0 and the number and percent of subjects with medical history will be summarized by (SOC) and Preferred Term (PT) for each treatment group based on the safety population.

### 7.9 Treatment Exposure

All exposure data will be listed by treatment, subject ID for safety population.

### 8 Intranasal Examination

Intranasal assessments collected at Screening (Visit 1) will be summarized by treatment group and laterality with counts and percentages.

### 9 Safety Analysis

The safety population will be used for all safety analyses. All recorded safety parameters will be listed by treatment, subject ID and date.

### 9.1 Adverse Events





The investigator will promptly review each Adverse Event (AE) for accuracy and completeness, and classify each AE according to its intensity, its relationship to study drug or administration procedure, and its seriousness. AEs will be coded using version 22.0 of the MedDRA dictionary. AEs will be monitored throughout the study and documented on the appropriate AE form. AEs will be categorized as ocular and non-ocular events as well as by system organ class (SOC) and preferred term (PT), seriousness, severity, and relation to study medications.

All treatment-emergent adverse events (TEAEs) will be summarized. A TEAE is defined as an AE that is new or worsened in severity compared to the first dose of study drug. All AEs will be presented in data listing with a flag indicating the event is a TEAE.

TEAEs will be summarized by subject. In addition, the number of TEAE episodes that occurred during the study will be provided in the overall summary of AE table.

The following presentations of TEAEs will be generated:

- Overall adverse events summary;
- Serious adverse events (SAE) by SOC and PT;
- TEAEs by Severity;
- TEAEs by Relationship;
- Ocular TEAEs by SOC and PT;
- Non-ocular TEAEs by SOC and PT;
- TEAEs leading to study discontinuation.

### 9.2 Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO DD version B3, March 2019) and summarized for each treatment group in the safety population. A prior medication is defined as any medication taken within 60 days before dosing on Day 1 in the study. Any medication taken from the day of first dose of the study treatment up to the day of last date of the study will be considered as a concomitant medication for analysis.

Table 1 describes the classification of prior and concomitant medications.









### Appendix 1 Schedule of Visits and Measurements

| Procedure | Screening (Visit 1) | Treatment a | 2 2 |
|---|---|---|---|
| | ` ′ | Pre-Treatment | Post-Treatment |
| Informed consent/HIPAA | X | | |
| Demographics | X | | |
| Medical history, prior medication(s), ocular history and updates | X | | |
| Eligibility criteria | X | | |
| Urine pregnancy test <sup>1</sup> | X <sub>1</sub> | | |
| OSDI© questionnaire | X | | |
| Eye Dryness Score (EDS) | X | | |
| Imaging of Goblet Cells with Heidelberg Retinal Tomograph 3® | | X | X |
| Imaging of Meibomian Glands with Oculus Keratograph 5M® | | X | X |
| Slit lamp biomicroscopy | X | X | |
| Corneal fluorescein staining | X | | |
| Schirmer's test | X | | |
| Schirmer's test with cotton swab stimulation | X | | |
| Intranasal examination | X | | |
| Randomization | | X | |
| Dispense investigational drug / placebo | | X | |
| Administer investigational drug / placebo | | | X |
| Concomitant medication | X | X | |
| AE Query | X | X | X |
| 1- If applicable for women of childbearing potential | | | |





### Appendix 2 Table of Contents

Table 14.1.1 Subjects Screened and Screen Failures (All Subjects)

 Table 14.1.2 Subject Disposition (All Subjects)

 Table 14.1.3 Demographics (Safety Population)

Table 14.1.4 Important Protocol Deviation (Safety Population)

 Fable 14.1.5.1 Ocular Medical History (Safety Population)

Fable 14.1.5.2 Non-Ocular Medical History (Safety Population)

able 14.1.6.1 Ocular Prior Medications (Safety Population)

Table 14.1.6.2 Non-Ocular Prior Medications (Safety Population)

Table 14.1.6.3 Ocular Concomitant Medications (Safety Population)

 Table 14.1.6.4 Non-Ocular Concomitant Medications (Safety Population)

Table 14.3.1 Overall Summary of Treatment-Emergent Adverse Events (Safety Population)

Fable 14.3.2.1 Ocular Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

able 14.3.2.2 Non-Ocular Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

able 14.3.3.1 Treatment-Emergent Adverse Events by Severity (Safety Population)

Table 14.3.3.2 Treatment-Emergent Adverse Events by Relationship (Safety Population)

Table 14.3.4 Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

 Table 14.3.5 Serious Treatment-Emergent Adverse Events Related to Study Drug (Safety Population)

Fable 14.3.6 Treatment-Emergent Adverse Events Leading to Study Discontinuation (Safety Population)

able 14.4.1 Intranasal Examination Results (Safety Population)

Listing 16.2.1 Demographics (All Subjects)

Listing 16.2.2 Subject Disposition at End of Study (All Population)

Listing 16.2.3 Protocol Deviations (Safety Population)

Listing 16.2.4 Inclusion/Exclusion Criterion Not Met (All Subjects)

Listing 16.2.5 Study Drug Exposure (Safety Population)

Listing 16.2.6 Prior and Concomitant Medications (Safety Population)

Listing 16.2.7 Medical History (Safety Population)





Listing 16.2.8 Intranasal Examination (Safety Population)
Listing 16.2.9 Treatment-Emergent Adverse Events (Safety Population)





### Appendix 3 Tableshell

Table 14.1.1 Subjects Screened and Screen Failures (All Subjects)

| | Table 14.1.1 |
|---|---|
| 8 | Subjects Screened and Screen Failures |
| | All Subjects |
| | N=XX |
| Category | n (%) |
| Number of subjects screened | XX |
| Number of subjects with screen failure | XX (XX.X) |
| Screen failure reason | |
| Non-Fatal Adverse Event | XX (XX.X) |
| Protocol Violation | XX (XX.X) |
| Lost to Followup | XX (XX.X) |
| Pregnancy | (X:XX) XX |
| Physician Decision | (X:XX) XX |
| Subject non-compliance | (X:XX) XX |
| Death | (X:XX) XX |
| Study Terminated by Sponsor | (X:XX) XX |
| Withdraw by Subject | (X:XX) XX |
| Other | XX (XX.X) |

O:\projects\ Oyster Point Pharma\OPP-005\tables\xxx.sas (ddmmmyyyy hh:mm) Source: Listings 16....





Table 14.1.2 Subject Disposition (All Subjects)

| | | | | | | | | | _ | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Total | N=xx | n (%) | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | Placebo | N=xx | n (%) | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <b>Table 14.1.2</b> | Subject Disposition<br>All Subjects | OC-01 1.2 mg/mL | N=xx | n (%) | XX | xx (xx.x) | xx (xx.x) | xx (xx.x) | | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | | | | Category | Randomized | Safety population [1] | Subjects completed study | Subjects discontinued from study (for reasons | other than study completion) | Non-Fatal Adverse Event | Protocol Violation | Lost to Followup | Pregnancy | Physician Decision | Subject non-compliance | Death | Study Terminated by Sponsor | Withdraw by Subject | Other |

Percentages are calculated based on all randomized subjects. [1] The safety population will include all randomized subjects who received study drug at Visit 2.





Table 14.1.3 Demographics (Safety Population)

| | Table 14.1.3 Demographics Safety Population | u | |
|---|---|---|---|
| | OC-01 1.2 mg/mL | | Total |
| Category | N=xx | N=xx | N=xx |
| Age (Year) | | | |
| u | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Range (min, max) | XX, XX | XX, XX | XX, XX |
| Quartiles (25th, median, 75th) | XX.X, XX.X, XX.X | XX.X, XX.X, XX.X | XX.X, XX.X, XX.X |
| Sex, n (%) | | | |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | (x.xx) xx | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Reported | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race, n (%) | | | |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Native Hawaiian or other Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 71 | | (11 17 | |

SD: Standard Deviation.





Table 14.1.4 Important Protocol Deviation (Safety Population)

| | (x-xx) xx (x-xx) xx | Deviation $1>$ $xx(xx,x)$ $xx(xx,x)$ $xx(xx,x)$ $xx(xx,x)$ | | ests with at least one major protocol $xx(xx,x)$ $xx(xx,x)$ $xx(xx,x)$ $xx(xx,x)$ | n (%) | N=xx | g/mL Placebo | Safety Population | Total N=xx n (%) xx (xx,x) xx (xx,x) xx (xx,x) | | Table 14.1.4 Important Protocol Dev Safety Population OC-01 1.2 mg/mL N=xx n (%) xx (xx,x) xx (xx,x) xx (xx,x) | No. of subjects with at least one major protocol deviation <major 1="" deviation=""> <maior 2="" deviation=""></maior></major> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Safety Population OC-01 1.2 mg/mL Placebo N=xx n (%) n (%) n (%) xx (xx,x) xx (xx,x) | Safety Population OC-01 1.2 mg/mL Placebo N=xx n (%) n (%) n (%) xx (xx,x) xx (xx,x) | Safety Population OC-011.2 mg/mL Placebo N=xx n (%) n (%) n (%) n (%) n (xx,x) xx (xx,x) | Safety Population OC-01 1.2 mg/mL Placebo N=xx N=xx n (%) n (%) tocol xx (xx,x) xx (xx,x) | Placebo N=xx n (%) | Placebo N=xx | wlation Placebo Placebo | Safety Population | | | iation | Important Protocol Dev | |
| Important Protocol Deviation Safety Population OC-01 1.2 mg/mL N=xx n (%) n (%) n (%) n (%) n (%) xx (xx,x) xx (xx,x | Important Protocol Deviation Safety Population Safety Population OC-01 1.2 mg/mL N=xx n (%) n (%) n (%) xx (xx,x) xx ( | Important Protocol Deviation Safety Population OC-01 1.2 mg/mL N=xx n (%) n (%) | Important Protocol Deviation Safety Population OC-01 1.2 mg/mL N=xx N=xx n (%) n (%) tocol xx (xx,x) xx (xx,x) | col Deviation ulation Placebo N=xx n (%) | col Deviation ulation Placebo N=xx | col Deviation ulation Placebo | Important Protocol Deviation<br>Safety Population | Important Protocol Deviation | | | Table 14.1.4 | |

Percentages are based on the total number of subjects in the Safety Analysis Set. Some subjects may have multiple major protocol deviations.





Table 14.1.5.1 Ocular Medical History (Safety Population)

| | Table 14.1.5.1 | | |
|---|---|---|---|
| | Ocular Medical History | ıry | |
| | Safety Population | | |
| | OC-01 1.2 mg/mL | Placebo | Total |
| MedDRA System Organ Class | N=xx | N=xx | N=xx |
| Preferred term | n (%) | n (%) | n (%) |
| Subjects with any Ocular Medical History | xx (xx,x) | xx (xx,x) | xx (xx,x) |
| System Organ Class 1 | xx (xx,x) | xx (xx,x) | xx (xx,x) |
| Preferred Term 1 | xx (xx,x) | XX (XX,X) | xx (xx,x) |
| Preferred Term 2 | xx (xx,x) | XX (XX,X) | xx (xx,x) |
| •••• | | | |
| System Organ Class xx | xx (xx,x) | xx (xx,x) | xx (xx,x) |
| Preferred Term 1 | xx (xx,x) | XX (XX,X) | xx (xx,x) |
| Preferred Term 2 | xx (xx,x) | xx (xx,x) | xx (xx,x) |
| ***** | | | |

Note: Ocular medical history was coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 22.0. Only medical histories collected on the CRF form of Ocular History are included for the summary.

Each subject could only contribute once to each of the incidence rates, regardless of the number of occurrences.

Table 14.1.5.2 Non-Ocular Medical History (Safety Population)

Programming note: same format as Table 14.1.5.1





| | Table 14.1.6.1 | | |
|---|---|---|---|
| ) | Ocular Prior Medications<br>Safety Population | | |
| | OC-01 | Placeho | Total |
| WHO Drug ATC2 | X=N | N=XX | N=XX |
| WHO Drug ATC4 | n (%) | n (%) | n (%) |
| Subjects with Any Ocular Prior Medications | XX (XX,X) | XX (XX,X) | XX (XX,X) |
| ATC2 1 | XX (XX,X) | XX (XX,X) | xx (xx,x) |
| ATC4 1 | xx (xx,x) | XX (XX,X) | xx(xx,x) |
| ATC4 2 | xx (xx,x) | XX (XX,X) | xx(xx,x) |
| ATC2 xx | xx (xx,x) | XX (XX,X) | xx(xx,x) |
| ATC4 1 | xx (xx,x) | XX (XX,X) | xx(xx,x) |
| ATC4 2 | xx(xx,x) | xx (xx,x) | xx(xx,x) |

A prior medication is defined as any medication taken within 60 days before dosing on Day 1. Each subject could only contribute once to each of the incidence Note: World Health Organization Drug Dictionary (WHO-DD) version WHODRUG GLOBAL B3 March 1, 2019 was used for medication coding. rates, regardless of the number of occurrences.





## Table 14.1.6.2 Non-Ocular Prior Medications (Safety Population)

Programming note: same format as Table 14.1.6.1.

## Table 14.1.6.3 Ocular Concomitant Medications (Safety Population)

Programming note: same format as Table 14.1.6.1.

ootnote

World Health Organization Drug Dictionary (WHO-DD) version WHODRUG GLOBAL B3 March 1, 2019 was used for medication coding. Concomitant medications are all medications taken from the day of first dose of the study treatment up to the day of last date of the study.

# Table 14.1.6.4 Non-Ocular Concomitant Medications (Safety Population)

Programming note: same format as Table 14.1.6.1.

Footnote

World Health Organization Drug Dictionary (WHO-DD) version WHODRUG GLOBAL B3 March 1, 2019 was used for medication coding. Concomitant medications are all medications taken from the day of first dose of the study treatment up to the day of last date of the study.





Table 14.3.1 Overall Summary of Treatment-Emergent Adverse Events (Safety Population)

| Overall Sun | Table 14.3.1<br>Overall Summary of Treatment-Emergent Adverse Events<br>Safety Population | nt Adverse Events | |
|---|---|---|---|
| | OC-01 1.2 mg/mL | Placebo<br>N=xx | Total |
| Category | n (%) | (%) u | n (%) |
| Subjects with any TEAE | xx (xx.x) | (x·xx) xx | (x.xx) xx |
| Subjects with any ocular TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any resolved ocular TEAEs | (x:xx) xx | (x·xx) xx | (x:xx) xx |
| Subjects with any non-ocular TEAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any treatment-emergent SAEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any treatment-related treatment | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any TEAE by maximum severity [1] | | | |
| Mild | xx (xx.x) | (x:xx) xx | xx (xx.x) |
| Moderate | xx (xx.x) | (x·xx) xx | (x:xx) xx |
| Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any TEAEs related to study drug | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects with any TEAEs related to study discontinuation | xx (xx.x) | (x·xx) xx | (x.xx) xx |
| Subjects with any TEAEs leading to death | xx (xx.x) | xx (xx.x) | xx (xx.x) |

[1] Subjects reporting more than one event are counted only once at the maximum severity reported.





| | | 4.3.2.1 | Table 14.3.2.1 |
|---|---|---|---|
| Ocular Trea | itment-Emergent Adverse Events by Syste<br>Safety Population | Ocular Treatment-Emergent Adverse Events by System Organ Class and Preferred Term<br>Safety Population | red Term |
| | OC-01 1.2 mg/mL | Placebo | Total |
| System Organ Class (SOC) | N=xx | N=xx | N=xx |
| Preferred Term (PT) | n (%) | n (%) | n (%) |
| Any Ocular TEAEs | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| System Organ Class xx | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | (x·xx) xx | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n (%) = number (percent) of subjects with events.

Note: A TEAE is defined as AE that is new or worsened in severity compared to the first dose of study drug. TEAEs were coded using MedDRA version 22.0.

### Table 14.3.2.2 Non-Ocular Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

Programming note: same format as Table 14.3.2.1.





Table 14.3.3.1 Treatment-Emergent Adverse Events by Severity (Safety Population)

| | | Table 14.3.3.1 | 3.1 | |
|---|---|---|---|---|
| | | Treatment-Emergent Adverse Events by Severity<br>Safety Population | e Events by Severity<br>tion | |
| | | OC-01 1.2 mg/mL | Placebo | Total |
| System Organ Class | | N=xx | N=xx | N=xx |
| Preferred Term | Severity | n (%) | n (%) | n (%) |
| Any TEAEs | Mild | XX (XX.X) | XX (XX.X) | xx(xx.x) |
| | Moderate | XX (XX.X) | XX (XX.X) | XX(XX.X) |
| | Severe | XX(XX.X) | XX (XX.X) | XX(XX.X) |
| System Organ Class 1 | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | XX (XX.X) | XX (XX.X) | xx(xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | Mild | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | Moderate | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | Severe | xx (xx.x) | xx (xx.x) | xx (xx.x) |

n (%) = number (percent) of subjects with events. Note: A TEAE is defined as AE that is new or worsened in severity compared to the first dose of study drug. TEAEs were coded using MedDRA version 22.0. [1] Subjects reporting more than one event are counted only once at the maximum severity reported.





Table 14.3.3.2 Treatment-Emergent Adverse Events by Relationship (Safety Population)

Programming note: same format as Table 14.3.3.1. Please change Severity to Relationship. The category of relationship includes Related, and Not Related.

Table 14.3.4 Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population) Programming note: same format as Table 14.3.2.1.

Table 14.3.5 Serious Treatment-Emergent Adverse Events Related to Study Drug (Safety Population)

Programming note: same format as Table 14.3.2.1.

Table 14.3.6 Treatment-Emergent Adverse Events Leading to Study Discontinuation (Safety Population) Programming note: same format as Table 14.3.2.1.





Table 14.4.1 Intranasal Examination Results (Safety Population)

| Table 14.4.1 | | Placebo | N=xx | 11/11 (%) | Left Nostril Right Nostril | | xx/xx $(xx.x)$ $xx/xx$ $(xx.x)$ | xx/xx $(xx.x)$ $xx/xx$ $(xx.x)$ |
|---|---|---|---|---|---|---|---|---|
| | Intranasal Examination Results<br>Safety Population | g/n | N=xx | n/N1 (%) | Right Nostril | | (x·xx) xx/xx | (x·xx) xx/xx |
| | | OC-01 1 | ŻŹ | II/II | Left Nostril | | (x.x) xx/xx | (x.x) xx/xx |
| | | | | | Visit/Result | Visit 1 [1] | Normal | Abnormal |

Column header counts are the number of treated subjects.

N1 are the number of treated subjects with non-missing data at given visit.

[1] Screening visit





### Oyster Point Pharma, Inc.

**Clinical Protocol: OPP-005:** 

A Single-Center, Randomized, Controlled, Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation (The IMPERIAL Study)



### Abbreviated Statistical Analysis Plan Version 1.0

Prepared by

Date: February 14, 2020



| Author: |
|---|
| <b>Study OPP-005:</b> A Single-Center, Randomized, Controlled, Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Goblet Cell and Meibomian Gland Stimulation (The IMPERIAL Study) |
| Brief Summary of Analysis: |
| The sample size for the study is not based on statistical power calculation and sample size at the end of the study is relatively small. For this reason, |
| Meibography Analysis: |
| Descriptive statistics consisting of the number of subjects (n), mean, standard deviation, median ,25 <sup>th</sup> and 75 <sup>th</sup> percentiles, and minimum and maximum will be used to summarize each time point (Pre-Treatment, Post Treatment) as well as the Change from Pre-treatment. Pre-treatment and post-treatment in area and perimeter |
| 2. A summary analysis will also utilize descriptive statistics consisting of the number of subjects (n), mean, standard deviation, 25 <sup>th</sup> and 75 <sup>th</sup> percentiles, and minimum and maximum. |
| 3. A by subject listing for both area and perimeter will be provided containing each subjects meibography number of meibography reads (n), mean, standard deviation, 25 and 75 <sup>th</sup> percentiles, and minimum and maximum. These statistics will summarize the change from pre-treatment meibography read results for each subject by eye laterality and lid discretion. |

Date: February 14, 2020

### **Goblet Cell Analysis:**

| 1. | A change from Pre-treatment analysis will be performed, maintaining intrasubject, eye | e |
|---|---|---|
| | laterality independence for both the active 0.2% OC-01 treatment group as well as | |
| | placebo. Descriptive statistics consisting of the number of subjects (n), mean, standard | 1 |
| | deviation, median ,25 <sup>th</sup> and 75 <sup>th</sup> percentiles, and minimum and maximum will be used | to |
| | summarize each time point (Pre-Treatment, Post Treatment) as well as the overall | |
| | Change from Pre-treatment. | |
| | | _ |



3. A by subject listing for both area and perimeter will be provided containing each subjects Goblet Cell measurement results detailing the eye laterality for each time point.

number of Goblet Cell measurements (n), mean, standard deviation, 25 and 75 percentiles, and minimum and maximum. These statistics will summarize the change from pre-treatment Goblet Cell measurement results for each subject by eye laterality.